CLINICAL TRIAL: NCT04255992
Title: Short Term Cardiovascular Effects and Oxidative Status of Calcium and Vitamin D Supplementation of Postmenopausal Hypertensive Blacks Women in Sub Saharan Africa
Brief Title: Short Term Cardiovascular Effects and Oxidative Status of Calcium and Vitamin D Supplementation of Postmenopausal Hypertensive Blacks Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, CN NGANOU-GNINDJIO, MD, MSc, Dr, Principal investigator, Yaounde Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: calcium and vitamin D in HW
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hypertension; Postmenopausal Disorder
Keywords: Blood pressure; Oxidative status
MeSH Terms: conditions — Hypertension | interventions — S100 Calcium Binding Protein G

STUDY DESIGN:
Intervention Model Description: This study is a double blind, randomized, controlled parallel clinical trial conducted at the Yaounde central hospital, Cameroon
Who Masked: Participant, Investigator
Masking Description: The double-blind model is applied to the study. Only the adjudicator, responsible for the distribution of medication knew the different regimes. Calcium and Vitamin D/Calcium were packaged in boxes of identical appearance and labeled for each participant by name and number of the randomization program. The randomization and packaging of the drugs was done by an investigator who had no clinical involvement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium arm (Active Comparator): 1000 mg Calcium tablet per day at 8am (+/- 1 hour) was add to the usual treatment for each patient. Patients are followed-up for a period of 08 weeks.
  Interventions: Dietary Supplement: Calcium Arm
- Vitamin D/Calcium (Active Comparator): 1000 mg/800UI of VitaminD/Calcium tablet per day at 8am (+/- 1 hour) was add to the usual treatment for each patient. Patients are followed-up for a period of 08 weeks.
  Interventions: Dietary Supplement: Vitamin D/Calcium

INTERVENTIONS:
Dietary Supplement: Calcium Arm — 1000 mg Calcium tablet / day will be added to the usual treatment for each patient for a period of 8 weeks.
  Arms: Calcium arm
Dietary Supplement: Vitamin D/Calcium — 1000 mg/800UI of the association Vitamin D/Calcium tablet / day will be added to the usual treatment for each patient for a period of 8 weeks.
  Arms: Vitamin D/Calcium

SUMMARY:
This study aims to determine the effect of calcium and vitamin D supplementation on oxidative status and blood pressure profile of postmenopausal patients with high blood pressure in Yaoundé, Cameroon.

This study is a double-arm, double-blind, randomized and parallel clinical trial conducted at the Yaoundé Central Hospital

DETAILED DESCRIPTION:
Aim: to determine and compare the short term effect of calcium and vitamin D supplementation on oxidative status and blood pressure profile of postmenopausal patients with high blood pressure in Yaoundé, Cameroon.

Method: A double-arm, double-blind, randomized and parallel clinical trial conducted at the Yaoundé Central Hospital. Postmenopausal hypertensive blacks women who are taking taking antihypertensives drugs since 12 months,without diabetes mellitus or any inflammatory disease or hypercalcemia, are randomize into 2 groups. Depending on the group, the intervention consisted of the administration of Calcium 1000 mg daily or Vitamin D/Calcium 1000 mg/800 UI daily for 08 weeks. The endpoints were the nycthemeral blood pressure profile, pro oxidant marker (malondialdehyde) and anti-oxidant marker (Ferric reducing antioxidant).

Progress: Recruitment for this study was completed in May 2019 with 22 patients.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal hypertensive women since 12 months
* On a stable antihypertensive therapies (determined by the investigator) for at least 3 months with no classes changes.
* Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* Diabetes mellitus or inflammatory diseases
* Hypercalcemia,
* Side effects affecting life quality of patients (determined by the Data Safety Monitoring Board).
* Withdrawal of consent

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal hypertensive women
Enrollment: 22 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Change in nycthemeral blood pressure profile (mmHg) | 8 weeks
  Change in nycthemeral blood pressure profile from baseline to week 08. By using Arterial Blood Pressure Monitoring.

SECONDARY OUTCOMES:
Change in serum concentration of oxidant marker: malondialdehyde (micromol/l) | 8 weeks
  Change in concentration of oxidant marker from baseline to week 8. By spectrophotometer

OTHER OUTCOMES:
Change in serum concentration of anti-oxidant markers: Ferric reducing antioxidant Power (micromol) | 8 weeks
  Change in concentration of anti oxidant marker from baseline to week 8. By spectrophotometer

CONTACTS AND LOCATIONS:
Locations (1):
- Yaounde Central Hospital, Cardiology department, Yaoundé, Cameroon